CLINICAL TRIAL: NCT03215407
Title: The Comparative Study of Safety and Effectiveness of Intra-articular Injection of Tocilizumab and Compound Betamethasone in Rheumatoid Arthritis of the Knee
Brief Title: The Comparative Study of Intra-articular Injection of Tocilizumab and Compound Betamethasone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhu, Associated Prof. of Medicine, Deputy Director of Rheumatology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinaPLAGH(Intraarticular+TCZ)
Record Dates: First submitted 2017-06-22; First posted 2017-07-12 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis of Knee
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-articular Tocilizumab (Experimental): Tocilizumab, solution, 80mg intra-articular.
  Interventions: Drug: Intra-articular Tocilizumab
- Intra-articular Compound Betamethasone (Active Comparator): Compound betamethasone, solution, 14mg intra-articular
  Interventions: Drug: Intra-articular Compound Betamethasone

INTERVENTIONS:
Drug: Intra-articular Tocilizumab — Patients will be randomly chosen to be intra-articular injected of tocilizumab injection
  Arms: Intra-articular Tocilizumab
Drug: Intra-articular Compound Betamethasone — Patients will be randomly chosen to be intra-articular injected of compound betamethasone injection
  Arms: Intra-articular Compound Betamethasone

SUMMARY:
Aim: Comparing the efficacy and safety of intra-articular injection of tocilizumab and compound betamethasone.

Study design: A randomized, single-blind, parallel controlled and one center trial design.

Sample size: 60 cases. Study content: Patients who meet inclusive criteria will be randomly divided into tocilizumab group and compound betamethasone group. In the baseline period, the investigators will collect patients' general information, disease information, disease activity score, laboratory results and images of articular ultrasound. After 4 weeks of injection, patients will be asked to come back, and their disease information, disease activity score, laboratory results as well as images of articular ultrasound will be collected. Finally, these data will be sorted and analyzed.

Hypothesis: The efficacy and safety of intra-articular injection of tocilizumab is better than that of compound betamethasone.

DETAILED DESCRIPTION:
Aim: Comparing the efficacy and safety of intra-articular injection of tocilizumab and compound betamethasone.

Study design: A randomized, single-blind, parallel controlled and one center trial design, the study period is 4 weeks.

Sample size: 60 cases. Study content: Patients who meet inclusive criteria will be randomly divided into tocilizumab group and compound betamethasone group according to the random number table. In the baseline period, the investigators will collect patients' general information, disease information, disease activity score, laboratory results and images of articular ultrasound. After 4 weeks of injection, patients will be asked to come back, and their disease information, disease activity score, laboratory results as well as images of articular ultrasound will be collected. Finally, these data will be sorted and analyzed.

Index of effect evaluation: 1) Articular ultrasound, OMERACT-EULAR composite PDUS synovitis score will be used to evaluate the condition of articulation; 2) Disease activity score, DAS28-CRP, DAS28-ESR; 3) Health Assessment Questionnaire, HAQ; 4) Rheumatoid and arthritis outcome score, RAOS; 5) composite change index, CCI score; 6) diameter of knee joint; 7) knee flexion range.

Hypothesis: The efficacy and safety of intra-articular injection of tocilizumab is better than that of compound betamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-65 years
2. Patients must be diagnosed as rheumatoid arthritis according to the 2010 ACR classification diagnostic criteria for RA for at least 6 months.
3. Patients' knee is swelling or has effusion.
4. Patients have used the same dosage of DMARDs or biologics for at least 6 weeks and continue using the drug until the end of the study.
5. If patients are using glucocorticoid or NSAIDs, the dosage must be stabilized for at least 4 weeks and continue until the end of the study.
6. Patients must understand the aim and steps of this study, can come back for follow-up timely.

Exclusion Criteria:

1. Patients' knee is out of shape. X-ray shows a moderate or severe damage of subchondral bone, or joint space is less than 3 mm.
2. Patients have received intra-articular injection of glucocorticoid or TNFi, joint replacement, or synovectomy.
3. Patients is suffering from other autoimmune diseases or Spondyloarthritis.
4. The skin of knee is damaged severely.
5. Patients is suffering from pulmonary tuberculosis, or Chest X-ray shows lesion signs related to tuberculosis.
6. For the last 3 months, patients have participated in other new drug's clinical trial.
7. Other patients who have been thought not suitable for the study by researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-12-12 (Estimated); Study Completion 2018-03-03 (Estimated)

PRIMARY OUTCOMES:
change from OMERACT-EULAR composite PDUS synovitis score at 4 weeks | 0 and 4 weeks
  use articular ultrasound to explore the condition of knee and evaluate the condition of knee by OMERACT-EULAR composite PDUS synovitis score

SECONDARY OUTCOMES:
change from disease activity score at 4 weeks | 0 and 4 weeks
  DAS28-CRP, DAS28-ESR
change from Health Assessment Questionnaire at 4 weeks | 0 and 4 weeks
  HAQ
change from Rheumatoid and arthritis outcome score at 4 weeks | 0 and 4 weeks
  RAOS
change from composite change index at 4 weeks | 0 and 4 weeks
  CCI score
change from diameter of knee joint at 4 weeks | 0 and 4 weeks
  diameter of knee joint
change from knee flexion range at 4 weeks | 0 and 4 weeks
  knee flexion range